CLINICAL TRIAL: NCT00647413
Title: Cancer Prevention by Reducing Exposure to Environmental Tobacco Smoke at Home
Brief Title: Prevent Exposure to Tobacco Smoke at Home [Gesunde Atemluft zu Hause]
Acronym: GESA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Deutsche Krebshilfe e.V., Bonn (Germany), Dr. Kohlhuber
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Krebshilfe-107539; DM8-IESO02
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Smoking; Passive Smoking; Exposure to Environmental Smoke
Keywords: smoking; passive smoking; exposure to environmental smoke; home smoking ban; urinary cotinine
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): expert system intervention on smoking behaviour + feedback of a biomarker
  Interventions: Behavioral: bio-chemical feedback and expert system intervention ETS

INTERVENTIONS:
Behavioral: bio-chemical feedback and expert system intervention ETS — Urinary cotinien will be measured using urine collected from the infants diaper. It will be analysed and the result will be explained to the participant in a written letter approximately 2 weeks after the intervention.
  The intervention will also be a counselling session about the consequences of ETS to the infant. The counselling will be guided by the principles of motivational intervieweing and an expert system letter tailored to the data assessed will be send to the participants
  Other Names: motivational interviewing; expert system intervention; tailored feedback
  Arms: 2

SUMMARY:
Background: Infants are at risk for tobacco-attributable diseases by being exposed to environmental tobacco smoke (ETS). International literature has shown that a home smoking ban can reduce ETS. The purpose of this study is to examine whether a brief feedback about urinary cotinine in infants and a counselling session about the consequences of ETS leads to a reduction of ETS.

All families with children up to an age of three years in the study region will be contacted by mail and asked for participation in this study. They will be randomised into an intervention and one control group. The intervention group will receive a ETS counselling session and detailed analysis of urinary cotinine (a biomarker of ETS) at their home. They will further receive written feedback approx. 2 weeks later. The control group will be visited and will answer a questionnaire and will receive brochures about ETS. They will receive a standard analysis feedback of urinary cotinine. There will be oine further assessment/ visit 12 months later. The outcome of this study is an anlysis of urinary cotinine and smoking behaviour and changes in cotinine and smoking behaviour.

ELIGIBILITY:
Inclusion Criteria:

* born in 2005, 2006 or 2007,
* being exposed to environmental tobacco smoke at home by at least one parent, living in the study region of west pommerania

Exclusion Criteria:

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
exposure to environmental tobacco smoke | 6 months

SECONDARY OUTCOMES:
smoking behaviour | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich John, Prof. Dr., Study Director — Institut für Epidemiologie und Sozialmedizin, University of Greifswald; Jochen René Thyrian, PhD, Principal Investigator — Institut für Epidemiologie und Sozialmedizin
Locations (1):
- Institut für Epidemiologie und Sozialmedizin, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Ulbricht S, Gross S, Meyer C, Hannover W, Nauck M, John U. Reducing tobacco smoke exposure in children aged below 4 years - a randomized controlled trial. Prev Med. 2014 Dec;69:208-13. doi: 10.1016/j.ypmed.2014.10.016. Epub 2014 Oct 18. PMID 25456808